CLINICAL TRIAL: NCT02847845
Title: A Clinical Study About Improvement of Chronic Fatigue After Taking Red Ginseng
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eun Jung Kim (Other)
Responsible Party: Sponsor-Investigator, Eun Jung Kim, Assistant professor, DongGuk University
Organization: DongGuk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: B080017-KCT0001935
Record Dates: First submitted 2016-07-05; First posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Fatigue Syndrome
Keywords: chronic fatigue syndrome; idiopathic chronic fatigue; red ginseng; cortisol; anti-oxidant
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Red ginseng powder capsule (Experimental): People in this group take a red ginseng powder capsule.
  Interventions: Dietary Supplement: red ginseng powder capsule
- Placebo powder capsule (Placebo Comparator): People in this group take a placebo powder capsule.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: red ginseng powder capsule — usage : 3C bid ac 30min dose : total 3g for 1day drug administration : oral administration administration session : 6weeks
  Arms: Red ginseng powder capsule
Dietary Supplement: Placebo — Control (Placebo) : red ginseng powder capsule(placebo) usage : 3C bid ac 30min dose : total 3g for 1day drug administration : oral administration administration session : 6weeks
  Arms: Placebo powder capsule

SUMMARY:
The purpose of this study is to verify the efficacy of taking red ginseng for chronic fatigue patient.

DETAILED DESCRIPTION:
Verify the efficacy and safety after taking red ginseng for chronic fatigue syndrome or idiopathic chronic fatigue patient. They were verified through not only survey like VAS change about fatigue, fatigue severity scale, Chalder fatigue severity questionnaire, SRI-short form , BDI , ISI EQ-5D-5L, ginseng subjective symptoms questionnaire but also an anti-oxidant test and a salivary cortisol test after 6 weeks after taking red ginseng or placebo drugs.

ELIGIBILITY:
Inclusion Criteria:

1. At least 19 years of age, but below 65 years of age
2. A subject who appear repetitive or continuous fatigue of unknown cause.
3. A subject who has not abnormal findings of blood pressure, complete blood cell count(Hb, Hct, WBC, glucose), biochemical examination(AST, ALT, creatinine), thyroid gland function test(TSH, FT4), Urine test(Urine glucose, Urine protein), Chest X-ray, and ECG for causing fatigue
4. A subject who voluntarily agrees to participate and signs after listening to explanation for purpose and characteristic about this clinical trial

Exclusion Criteria:

1. A subject who has history or PI for chronic fatigue
2. A subject who takes this drug in 2 weeks : antidepressant drug, anti-anxiety drug,sleeping pill, an antihistamine etc.
3. Pregnant, lactating women or a subject who has plan pregnancy.
4. A subject who receive medical treatment or takes dietary supplement(vit B,C etc) for chronic fatigue in 2 weeks.
5. A subject who has night duty, shift work or heavy work
6. A subject who is judged as being not fit by a specialist

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
100mm visual analogue scale(VAS) about fatigue change | at 1(screening),2(baseline),3(after 2 weeks of administration), 4(after 4 weeks of administration), 5(after 6 weeks of administration) and 6(follow up evaluation after 10 weeks of administration) visit
  The patient is asked to indicate their perceived fatigue intensity along a 100 mm horizontal line, where '0' represents 'no fatigue' and '100', 'unbearable fatigue'

SECONDARY OUTCOMES:
fatigue severity scale change | at 2(baseline),3(after 2 weeks of administration), 4(after 4 weeks of administration), 5(after 6 weeks of administration) and 6(follow up evaluation after 10 weeks of administration) visit
  The FSS is a self-administered questionnaire with 9 items (questions) investigating the severity of fatigue in different situations during the past week. Grading of each item ranges from 1 to 7, where 1 indicates strong disagreement and 7 strong agreement, and the final score represents the mean value of the 9 items
Chalder fatigue severity questionnaire change | at 2(baseline),3(after 2 weeks of administration), 4(after 4 weeks of administration), 5(after 6 weeks of administration) and 6(follow up evaluation after 10 weeks of administration) visit
  The Chalder fatigue severity questionnaire is composed of 11 questions about fatigue. Grading of each item ranges from 0 to 9, where 0 indicate non-fatigue and 9 strong fatigue
a short form of stress response inventory,SRI-short form change | at 2(baseline),3(after 2 weeks of administration), 4(after 4 weeks of administration), 5(after 6 weeks of administration) and 6(follow up evaluation after 10 weeks of administration) visit
  SRI-short form is composed of 22 items about stress response. 22 items are classified into three categories(Somatization,anger and depression).
beck depression inventory, BDI change | at 2(baseline),5(after 6 weeks of administration) and 6(follow up evaluation after 10 weeks of administration) visit
  When the test is scored, a value of 0 to 3 is assigned for each answer and then the total score is compared to a key to determine the depression's severity.
insomnia severity index, ISI change | at 2(baseline),3(after 2 weeks of administration), 4(after 4 weeks of administration), 5(after 6 weeks of administration) and 6(follow up evaluation after 10 weeks of administration) visit
  The ISI is composed of seven items assessing recent problems with sleep onset, sleep maintenance and early morning awakening, interference of sleep problems with daily functioning and perceived prominence of impairment attributed to the sleep problem, concern about sleep problems and satisfaction with sleep patterns. Perceived severity of each item is rated on a 0-4 scale and a total score, which ranges from 0 to 28 obtains from summing the items ratings
EuroQol - 5 Dimensions - 5 Levels, EQ-5D-5L change | at 2(baseline),3(after 2 weeks of administration), 4(after 4 weeks of administration), 5(after 6 weeks of administration) and 6(follow up evaluation after 10 weeks of administration) visit
  The EuroQOL - 5 Dimensions (EQ-5D) was employed for measuring health-related quality of life. It consisted of a weighted sum of five dimensions: Mobility, Self-care, Usual activities, Pain/Discomfort and Anxiety/Depression, which provided a simple descriptive profile and a single index value for health status . We used a recently developed version, the EQ-5D-5L, which includes five-level response options: no problems, slight problems, moderate problems, severe problems, and extreme problems
derivatives of Reactive Oxygen Metabolites (d-ROMs) change | at 2(baseline) and 5(after 6 weeks of administration) visit
  measure antioxidant levels in blood
Biological Antioxidant Potential (BAP) change | at 2(baseline) and 5(after 6 weeks of administration) visit
  measure antioxidant levels in blood
Thiobarbituric Reactive Acid Substances(TBARs) change | at 2(baseline) and 5(after 6 weeks of administration) visit
  measure antioxidant levels in blood
Superoxide Dismutase(SOD) change | at 2(baseline) and 5(after 6 weeks of administration) visit
  measure antioxidant levels in blood
Stress hormone test | at 2(baseline) and 5(after 6 weeks of administration) visit
  measure cortisol level in saliva
  First saliva sample : 07:00-09:00 (within 30 minutes after waking up)
  Second saliva sample :
  11:00-13:00
  Third saliva sample :
  16:00-18:00
  fourth saliva sample : 22:00-00:00
ginseng subjective symptoms questionnaire change | at 2(baseline),3(after 2 weeks of administration), 4(after 4 weeks of administration) and 5(after 6 weeks of administration) visit
  ginseng subjective symptoms questionnaire is composed of 13 items about subjective symptoms after taking red ginseng
check abnormal responses | at 1(screening),2(baseline),3(after 2 weeks of administration), 4(after 4 weeks of administration), 5(after 6 weeks of administration) and 6(follow up evaluation after 10 weeks of administration) visit

CONTACTS AND LOCATIONS:
Overall Officials: Eun Jung Kim, Ph.D, Principal Investigator — DongGuk University
Locations (1):
- Dongguk university Bundang Oriental Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided